CLINICAL TRIAL: NCT00292838
Title: Relative Potency of Inhaled Corticosteroids: Validation of a Clinical Model
Brief Title: Relative Potency of Inhaled Corticosteroids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RP#01-1929
Record Dates: First submitted 2006-02-14; First posted 2006-02-16 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Eosinophilic bronchitis with asthma; Eosinophilic bronchitis without asthma
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

INTERVENTIONS:
Drug: fluticasone 25, 50, 100, 200 mcg

SUMMARY:
To investigate the validity of a clinical model to determine the relative potency of different preparations of inhaled corticosteroids used for the treatment of asthma or of eosinophilic bronchitis without asthma.

ELIGIBILITY:
Inclusion Criteria:

* Sputum eosinophilia >3%
* Adults age 18-70 years
* History of episodic wheeze, chest tightness, dyspnea or cough within the last 12 months.
* FEV1 ≥ 60% predicted
* Steroid naive or on not more than 500 µg a day of beclomethasone or equivalent.
* Able to give written informed consent

Exclusion Criteria:

1. Recent asthma or COPD exacerbation (as judged by the clinician) due to respiratory infection within the last month
2. Relevant seasonal allergen exposure within 4 weeks or within the course of the study
3. Treatment with prednisone or antibiotics or hospitalisation within the past 6 weeks
4. Other respiratory diseases
5. Women who are pregnant or unwilling to use appropriate contraception during the study
6. Unable to withhold short-acting ß-agonist treatment for 6 hours before visit

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2001-01; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Sputum eosinophils

SECONDARY OUTCOMES:
Exhaled nitric oxide, FEV1, FEF25-75%

CONTACTS AND LOCATIONS:
Overall Officials: Frederick E Hargreave, MD, Principal Investigator — McMaster University
Locations (1):
- Firestone Institute for Respiratory Health, St. Joseph's Healthcare, Hamilton, Ontario, Canada